CLINICAL TRIAL: NCT06793644
Title: Prospective Observational Study of ICG Fluorescence Imaging in Open Fracture and Infection Patients: Early Comparison With a Novel Imaging Device
Brief Title: Study of ICG Fluorescence Imaging in Open Fracture and Infection Patients
Acronym: cBPI
Status: Recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Section Chief Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02002551
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-01

CONDITIONS: Fractures, Bone; Trauma Injury
Keywords: Immunofluorescence; Orthopaedic Trauma; Infection
MeSH Terms: conditions — Fractures, Bone; Accidental Injuries; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Established SSI Fracture Cohort: Patients 18 years of age or older. Extremity fracture. Prior definitive fracture management with external fixation, internal fixation, or joint fusion. Superficial, deep, or organ space SSI (as per CDC criteria) at the fracture site that requires operative management. Will have all fracture care surgeries performed by a participating surgeon or delegate. Provision of informed consent
  Interventions: Drug: Immunofluorescence Imaging
- Open Fracture Cohort: Patients 18 years of age or older. Open extremity fracture. Planned definitive fracture management with external fixation, internal fixation, or joint fusion.
  Open fracture wound management that includes formal surgical debridement within 72 hours of their injury. Will have all planned fracture care surgeries performed by a participating surgeon or delegate. Provision of informed consent.
  Interventions: Drug: Immunofluorescence Imaging

INTERVENTIONS:
Drug: Immunofluorescence Imaging — Patients will be administered FDA approved ICG through intravenous injection and imaged by a FDA approved surgical microscope (Spy Elite) which is 0.5 meter away from the subject. Both ICG fluorescence and the two imaging systems have been used for routine clinical practice for many years. Figure (a) shows the Schematic sketch of the imaging systems. ICG fluorescence imaging utilizes intravenously injected ICG, which is a fluorescent dye that is FDA-approved for clinical use, illuminated with near-infrared light. The ICG dye is indirectly activated and the dynamic fluorescence due to bone perfusion can be captured by a video rate imaging system.

SUMMARY:
The purpose of this study is to determine whether an indocyanine green (ICG) fluorescence imaging system (cBPI) can be used to provide surgeons with information about bone health or bone blood flow. This will help surgeons better understand the healing potential of bone and relative risk of complication. This is important to help surgeons select the most appropriate treatment for severe traumatic injuries and infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Open extremity fracture, planning for management with external fixation, internal fixation or joint fusion.
* Fracture Related Infection, planning for management with debridement and possible removal of hardware.
* Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
* Provision of informed consent.

Exclusion Criteria:

* Inability of patient to provide informed consent
* Fracture of the hand.
* Iodine allergy.
* Burns at the fracture site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present with an open fracture or fracture related infection.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants who undergo an unplanned fracture-related reoperation | 12 Months
  All unplanned reoperations will be documented using a specific case report form
Number of participants who experience a post-procedure surgical site infection | 12 Months
  Post-procedure surgical site infection using Centers for Disease Control criteria will be documented at each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No